CLINICAL TRIAL: NCT06148714
Title: A Randomized-Controlled Trial to Examine the Effects of a Daily Probiotic Supplement on Common Symptoms of Menopause
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maneuver Marketing (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 20379
Record Dates: First submitted 2023-11-19; First posted 2023-11-28 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Menopause

STUDY DESIGN:
Intervention Model Description: Randomized-Controlled Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study will be triple-blinded in that the study participants, the study coordinators, and the data analysis team will be blinded to the intervention or product allocation. Only the sponsor will know which product contains the active ingredients. After the study analysis is complete, the allocation will be unblinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Provitalize Probiotic (Experimental): Participants will take 2 capsules every morning on an empty stomach before their first meal of the day.
  Interventions: Dietary Supplement: Provitalize Natural Menopause Probiotic
- Placebo (Placebo Comparator): Participants will take 2 capsules every morning on an empty stomach before their first meal of the day.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Provitalize Natural Menopause Probiotic — Supplement containing a Probiotic blend of Bifidobacterium breve, Lactobacillus Gasseri, and Bifidobacterium animalis subsp. Lactis.
  Arms: Provitalize Probiotic
Other: Placebo — Placebo comparator containing Pure hydroxypropyl methylcellulose (HPmC) with food dye.
  Arms: Placebo

SUMMARY:
Symptoms of menopause can significantly affect overall quality of life. It is hypothesized that probiotic supplements can reduce the severity of these symptoms. This 90-day randomized controlled trial will examine the effects of the Provitalize Natural Menopause Probiotic on weight loss, waist circumference, sleep, and symptoms of menopause including hot flashes, night sweats, mood swings, anxiety, fatigue and brain fog. Participants will take either the test product or a placebo daily. All participants will complete study-specific questionnaires and provide sleep data from their Fitbit at Baseline, Day 30, Day 60 and Day 90. At Baseline, Day 30, Day 60 and and Day 90, participants will also provide a bodyweight measurement and a waist circumference measurement.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 45-65 years old
* Must experience hot flashes and/or night sweats at least once per day
* Must also be experiencing at least two symptoms of menopause, such as sleep disturbances, mood changes, fatigue and lack of energy, changes in sexual function, urinary changes, weight gain, or vaginal changes
* Can be either natural or surgical menopause
* Has not had a period in the last 12 consecutive months
* Willing to adhere to the study protocol for the duration of the study
* Willing to stop taking any other herbal remedies or supplements for the duration of the study
* Self-reports as "generally healthy"
* Has never taken Provitalize before
* No planned invasive medical procedures for the duration of the study or in the three weeks leading up to the study start

Exclusion Criteria:

* Not experiencing hot flashes and/or night sweats at least once per day and two other symptoms of menopause such as sleep disturbances, mood changes, fatigue and lack of energy, changes in sexual function, urinary changes, irregular or absent periods, or vaginal changes
* Unwilling to stop taking any other herbal remedies or supplements for the duration of the study
* Current use of conventional hormone replacement therapies, or plan to start during the study duration
* Current use of hormonal birth control, or plan to start during the study duration
* Known allergies or hypersensitivities to any product ingredients
* Current or history of uterine fibroids, endometriosis, polycystic ovarian syndrome, or history of abnormal pap smear
* Anyone with any known severe allergies requiring the use of an epi-pen
* Unwilling to adhere to the study protocol
* Anyone living with uncontrolled or chronic health disorders, including oncological or psychiatric disorders
* Pregnant, breastfeeding or trying to conceive
* Currently taking a prescription sleep aid

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
Change in body weight. [Timeframe: Baseline to Day 90] | 90 days
  Participants will weigh themselves using a Fitbit Smart Scale that they will be provided with.
Change in waist circumference. [Timeframe: Baseline to Day 90] | 90 days
  Participants will measure their waist circumference using a tape measure that they will be provided with.
Changes in scores on the Bristol Stool Chart. [Timeframe: Baseline to Day 90] | 90 days
  The Bristol Stool Chart is widely used as a research tool to evaluate the effectiveness of treatments for various diseases of the bowel. Types 1 and 2 indicate constipation, with 3 and 4 being the ideal stools as they are easy to defecate while not containing excess liquid, 5 indicating lack of dietary fiber, and 6 and 7 indicate diarrhoea.

SECONDARY OUTCOMES:
Changes in the frequency of hot flashes. [Timeframe: Baseline to Day 90] | 90 days
  Measured via study-specific questionnaires using a 5-point Likert scale. A lower score indicates a more favourable response, with 0=Not noticeable and 4=Severe.
Changes in the frequency of night sweats. [Timeframe: Baseline to Day 90] | 90 days
  Measured via study-specific questionnaires using a 5-point Likert scale. A lower score indicates a more favourable response, with 0=Not noticeable and 4=Severe.
Changes in the severity of brain fog experienced. [Timeframe: Baseline to Day 90] | 90 days
  Measured via study-specific questionnaires using a 5-point Likert scale. A lower score indicates a more favourable response, with 0=Not noticeable and 4=Severe.
Changes in the severity of mood swings. [Timeframe: Baseline to Day 90] | 90 days
  Measured via study-specific questionnaires using a 5-point Likert scale. A lower score indicates a more favourable response, with 0=Not noticeable and 4=Severe.
Changes in the severity of fatigue. [Timeframe: Baseline to Day 90] | 90 days
  Measured via study-specific questionnaires using a 5-point Likert scale. A lower score indicates a more favourable response, with 0=Not noticeable and 4=Severe.
Changes in the severity of bloating. [Timeframe: Baseline to Day 90] | 90 days
  Measured via study-specific questionnaires using a 5-point Likert scale. A lower score indicates a more favourable response, with 0=Not noticeable and 4=Severe.
Changes in the frequency of bloating. [Timeframe: Baseline to Day 90] | 90 days
  Measured via study-specific questionnaires using a 5-point Likert scale. A lower score indicates a more favourable response, with 0=Not noticeable and 4=Severe.
Changes in the severity of joint pain. [Timeframe: Baseline to Day 90] | 90 days
  Measured via study-specific questionnaires using a 5-point Likert scale. A lower score indicates a more favourable response, with 0=Not noticeable and 4=Severe.
Changes in total time asleep. [Timeframe: Baseline to Day 90] | 90 days
  Measured using Fitbit wearable sleep tracker.
Changes in overall sleep score provided by Fitbit wearable sleep tracker. [Timeframe: Baseline to Day 90] | 90 days
  The sleep score is based on heart rate, the time spent awake or restless, and sleep stages. The score is given out of 100, with 100 indicating the best possible score.
Changes in total time awake at night. [Timeframe: Baseline to Day 90] | 90 days
  Measured using Fitbit wearable sleep tracker.

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: Undecided